CLINICAL TRIAL: NCT05146739
Title: A Phase 1 and Pharmacokinetic Study of Uproleselan (GMI-1271, NSC #801708) in Combination With Fludarabine and Cytarabine for Patients With Acute Myeloid Leukemia, Myelodysplastic Syndrome or Mixed Phenotype Acute Leukemia That Expresses E-selectin Ligand on the Cell Membrane and is in Second or Greater Relapse or That is Refractory to Relapse Therapy
Brief Title: Highest Dose of Uproleselan in Combination With Fludarabine and Cytarabine for Patients With Acute Myeloid Leukemia, Myelodysplastic Syndrome, or Mixed Phenotype Acute Leukemia Relapsed or Refractory That Expresses E-selectin Ligand on the Cell Membrane
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Children's Oncology Group (Network); LLS PedAL LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-10020; NCI-2021-10020 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEPN2113-APAL2020C; PEPN2113 (Other: Pediatric Early Phase Clinical Trial Network); PEPN2113 (Other: CTEP); UM1CA228823 (NIH)
Record Dates: First submitted 2021-11-18; First posted 2021-12-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia Post Cytotoxic Therapy; Myelodysplastic Syndrome Post Cytotoxic Therapy; Myeloid Leukemia Associated With Down Syndrome; Recurrent Acute Myeloid Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Mixed Phenotype Acute Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes | interventions — Cytarabine; fludarabine; Leucovorin; uproleselan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (uproleselan, fludarabine, cytarabine) (Experimental): Patients receive uproleselan IV QD over 20 minutes on day 1 and IV over 20 minutes BID on days 2-8, fludarabine IV QD over 30 minutes on days 2-6, and high dose cytarabine IV QD over 1-3 hours on days 2-6. Patients also receive cytarabine IT on day 0 then weekly starting on day 7-28 or ITT on day 0 then weekly starting on day 7-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with Down syndrome will receive leucovorin PO or IV BID following each intrathecal administration of methotrexate.
  Interventions: Drug: Cytarabine; Drug: Fludarabine; Drug: Leucovorin; Drug: Triple Intrathecal Chemotherapy; Drug: Uproleselan

INTERVENTIONS:
Drug: Cytarabine — Given IV and IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Leucovorin — Give PO or IV
  Other Names: Folinic acid
Drug: Triple Intrathecal Chemotherapy — Given IT
  Other Names: Triple Combination IT Chemotherapy; Triple IT Chemotherapy
Drug: Uproleselan — Given IV
  Other Names: GMI-1271

SUMMARY:
This phase I trial tests the safety, side effects, and determination of the best dose of uproleselan in combination with fludarabine and cytarabine in treating patients with acute myeloid leukemia, myelodysplastic syndrome or mixed phenotype acute leukemia that has come back (relapsed) or does not respond to treatment (refractory) and that expresses E-selectin ligand on the cell membrane. Uproleselan binds to E-selectin expressed on endothelial cells of the bone marrow and prevents their interaction with selectin-E ligand-expressing cancer cells. This may prevent leukemia cells from being sequestered in the bone marrow niche and escaping the effect of chemotherapy. Chemotherapy drugs, such as fludarabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving uproleselan in combination with fludarabine and cytarabine may expose more cancer cells to the effect of chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose or recommended Phase 2 dose of uproleselan (GMI-1271) administered in combination with fludarabine and cytarabine to patients with acute myeloid leukemia (AML), myelodysplastic syndrome (MDS) or mixed phenotype acute leukemia (MPAL) whose blasts express the E-selectin ligand and that are in second or greater relapse or refractory to relapse therapy.

II. To characterize the pharmacokinetics of uproleselan (GMI-1271) in combination with fludarabine and cytarabine in patients with refractory and/or relapsed AML, MDS or MPAL.

III. To define and describe the toxicities of uproleselan (GMI-1271) in combination with fludarabine and cytarabine among patients with relapsed and/or refractory AML, MDS or MPAL.

SECONDARY OBJECTIVES:

I. To describe the expression of E-selectin ligand on the surface of myeloid leukemic blasts at relapse prior to initiation of uproleselan (GMI-1271) in combination with fludarabine and cytarabine and at completion of the cycle.

II. To describe the antileukemic activity of uproleselan (GMI-1271) (Children's Oncology Group [COG]-complete remission [CR]/CR with partial recover of platelet count [CRp]/CR with incomplete blood count recovery [CRi] and rates of minimal residual disease [MRD] negative response after up to two cycles of therapy) in combination with fludarabine and cytarabine within the limits of a Phase 1 study.

EXPLORATORY OBJECTIVE:

I. To determine the largest relative reduction in myeloid leukemic blast percentage in the bone marrow, calculated from baseline at time of enrollment to up to two cycles of therapy.

OUTLINE: This is a dose escalation study of uproleselan.

Patients receive uproleselan intravenously (IV) once daily (QD) over 20 minutes on day 1 and IV over 20 minutes twice daily (BID) on days 2-8, fludarabine IV QD over 30 minutes on days 2-6, and high dose cytarabine IV QD over 1-3 hours on days 2-6. Patients also receive cytarabine intrathecal therapy (IT) or intrathecal triple therapy (ITT) on day 0. CNS2 and CNS3 patients receive additional cytarabine IT or ITT once weekly starting on day 7-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with Down syndrome will receive leucovorin orally (PO) or IV BID following each intrathecal administration of methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be enrolled on APAL2020SC (NCT04726241)-Pediatric Acute Leukemia (PedAL) Screening Trial - Developing New Therapies for Relapsed Leukemias - A Leukemia & Lymphoma Society and COG Groupwide Screening Protocol
* Patients must be >= 1 year and <18 years of age at the time of study enrollment
* Patients, with or without Down syndrome (DS), and with de novo acute myeloid leukemia, therapy-related acute myeloid leukemia, myelodysplastic syndrome with increased blasts (MDS-IB), therapy-related myelodysplastic syndrome with increased blasts (MDS-IB) or mixed phenotype acute leukemia that expresses E-selectin ligand on the cell membrane according to APAL2020SC screening results and meet one of the following:

  * Second or greater relapse or refractory AML as defined below, including isolated extramedullary disease (EMD), but excluding isolated central nervous system (CNS) or isolated testicular disease.
  * Second or greater relapse or refractory myelodysplastic syndrome (MDS) with increased blasts (MDS-IB).
  * Second or greater relapse or refractory mixed phenotype acute leukemia (MPAL)

    * Note: Documentation of E-selectin expression by multidimensional flow cytometry (MDF) at the central laboratory (Hematologics, Inc.) on the most recent bone marrow sample prior to the diagnosis of the current relapsed or refractory disease is acceptable for eligibility to this study in the event of isolated extramedullary disease, inability to obtain a bone marrow aspirate or lack of leukemic blasts in the peripheral blood
* Bone marrow relapse and MDF - MRD relapse: (patients must meet one of the following criteria to be defined as having relapse disease)

  * A single bone marrow sample showing >= 1% leukemic blasts by multidimensional flow cytometry performed at the central laboratory (performed only at Hematalogics through the screening study APAL2020SC).
  * In cases where a bone marrow aspirate cannot be obtained because of extensive fibrosis, blast count can be obtained from touch imprints or estimated from an adequate bone marrow core biopsy. A complete blood count documenting the presence of at least 1,000/ uL (i.e., a white blood count [WBC] count >= 10,000/uL with >= 10% blasts or a WBC count of >= 5,000/uL with >= 20% blasts) circulating leukemic cells (blasts) can also be used if a bone marrow aspirate or biopsy cannot be performed
* Extramedullary relapse: Biopsy proven extramedullary disease after documented complete remission
* Refractory disease and MDF - MRD refractory: Following a re-induction cycle after any relapse, presence of >= 1% leukemic blasts by multidimensional flow cytometry performed at the central laboratory (performed only at Hematologics through the screening study APAL2020SC), OR there is persistent extramedullary disease. In cases where a bone marrow aspirate cannot be obtained because of extensive fibrosis, assessment of refractory disease will be defined as described
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50 for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age. Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have fully recovered (grade <2) from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, eg, blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive:

    * >= 14 days must have elapsed after the completion of other cytotoxic therapy, with the exception of hydroxyurea
    * NOTE: Cytoreduction with hydroxyurea must be discontinued >= 24 hours prior to the start of protocol therapy
  * Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total-body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Patients must be off calcineurin inhibitors for at least 28 days prior to the start of protocol therapy. Patients may be on physiological doses of steroids (equivalent to =<10 mg prednisone daily for patients >=18 years or =<10mg/m2/day for patients <18years)
    * Autologous stem cell infusion including boost infusion: >= 30 days
  * Cellular Therapy: >= 30 days after the completion of any type of cellular therapy (eg, modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * External beam radiation therapy (XRT)/External Beam Irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
  * Patients must not have received prior exposure to uproleselan (GMI-1271). NOTE: Prior therapy with fludarabine and/or cytarabine is permitted
* For patients with leukemia:

  * Platelet count >= 25,000/uL (may receive platelet transfusions)
* Estimated glomerular filtration rate (eGFR) >= 70 mL/min/1.73 m^2

  * "Bedside" Schwartz formula (2009): eGFR = 0.413 x (height [cm] /serum creatinine [mg/dL]) OR
  * Measured GFR >= 70 mL/min/1.73 m^2. If measured GFR is used, it must be performed using direct measurement with a nuclear blood sampling method or small molecule clearance method (iothalamate or other molecule per institutional standard).
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 3x ULN (unless attributed to leukemic involvement)
* Albumin >= 2 g/dL
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study

Exclusion Criteria:

* Patients with any of the following diagnoses

  * Patients with isolated relapsed or refractory central nervous system (CNS) disease or isolated relapsed or refractory testicular disease
  * Patients with acute promyelocytic leukemia (APL)
  * Patients with juvenile myelomonocytic leukemia (JMML)
  * Patients with a known congenital bone marrow failure syndrome
* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies, OR because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (e.g., male or female condom) for the duration of the study and for 3 months after the last dose of uproleselan (GMI-1271). Abstinence is an acceptable method of birth control
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible except patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-05-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of uproleselan | Up to 28 days
  The MTD/RP2D will be the maximum dose at which fewer than one-third of patients experience dose limiting toxicities.
Cycle 1 dose limiting toxicity of uproleselan | Up to 28 days
  The frequency (%) of patients who experience a dose limiting toxicity on cycle 1, stratified by study part and dose level.
Area under the plasma concentration versus time curve of uproleselan | Up to 6 days
  The median (min, max) of the area under the plasma concentration versus time curve of uproleselan will be assessed immediately pre-dose as well as 30 minutes, 1 hour, 2 hour, and 4-hours post-dose on day 1 and day 6 of cycle 1, stratified by study part and dose level. Patients who weigh < 10 kilograms will have a 1.5 hour post-dose sample instead of the 1 hour and 2 hour post-dose samples.
Total plasma clearance of uproleselan | Up to 6 days
  The median (min, max) of the total plasma clearance of uproleselan will be assessed immediately pre-dose as well as 30 minutes, 1 hour, 2 hour, and 4-hours post-dose on day 1 and day 6 of cycle 1, stratified by study part and dose level. Patients who weigh < 10 kilograms will have a 1.5 hour post-dose sample instead of the 1 hour and 2 hour post-dose samples.
Elimination half-life of uproleselan | Up to 6 days
  The median (min, max) of the elimination half-life of uproleselan will be assessed immediately pre-dose as well as 30 minutes, 1 hour, 2 hour, and 4-hours post-dose on day 1 and day 6 of cycle 1, stratified by study part and dose level. Patients who weigh < 10 kilograms will have a 1.5 hour post-dose sample instead of the 1 hour and 2 hour post-dose samples.
Maximum concentration of uproleselan | Up to 6 days
  The median (min, max) of the maximum concentration of uproleselan will be assessed immediately pre-dose as well as 30 minutes, 1 hour, 2 hour, and 4-hours post-dose on day 1 and day 6 of cycle 1, stratified by study part and dose level. Patients who weigh < 10 kilograms will have a 1.5 hour post-dose sample instead of the 1 hour and 2 hour post-dose samples.

SECONDARY OUTCOMES:
Expression of E-selectin ligand on the surface of myeloid leukemic blasts of uproleselan | Up to 28 days
  Frequency (%) of subjects with positive expression of E-selectin ligand defined as an expression level above twice the native autofluorescence in 30% of myeloid blasts prior to initiation of uproleselan and at completion of cycle 1 stratified by study part and dose level.
Antileukemic activity of uproleselan | Up to 56 days
  Frequency (%) of subjects who respond to therapy defined as minimal residual disease negative if < 5% blasts at enrollment or complete remission (CR)/CR with partial recover of platelet count/CR with incomplete blood count recovery (attaining < 5% blasts, no evidence of circulating leukemic blasts or extramedullary disease and recovery of peripheral blood counts) if at least 5% blasts at enrollment stratified by study part and dose level.

OTHER OUTCOMES:
Relative reduction in myeloid leukemic blast percentage in bone marrow of uproleselen | Up to 56 days
  Median (min, max) percent change in myeloid leukemic blasts in bone marrow after 2 cycles of therapy versus baseline stratified by study part and dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Sulis, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (19):
- United States (19):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05146739/ICF_000.pdf